CLINICAL TRIAL: NCT00991237
Title: Pulsed Radiofrequency Treatment of the Lumbar Dorsal Root Ganglion for Patients With Chronic Lumbosacral Radicular Pain
Brief Title: PRF Treatment for Patients With Chronic Lumbosacral Radicular Pain Compared to Conventional Medical Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other); Sint Jozef Hospital Bornem en Willebroek Belgium (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NL28367.068.09
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Lumbosacral Radicular Syndrome
Keywords: NRS; GPE; pain reduction; quality of life
MeSH Terms: interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pain reduction (Experimental)
  Interventions: Other: Pulsed Radiofrequency

INTERVENTIONS:
Other: Pulsed Radiofrequency — Pulsed Radiofrequency
  Other Names: PRF

SUMMARY:
The purpose of the study is to evaluate the effect of PRF treatment adjacent to the lumbar dorsal root ganglion (DRG) of L5 or S1 in patients with a chronic lumbosacral radicular syndrome (LRS).

Prospective, single blinded, multicenter clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms more than 3 months 18,48
* Optimized conventional medical management at least for 1 month
* Pain radiating into the leg, up to the hallux (big toe) (L5) or little toe (S1)
* The pain in the leg dominates over a possible lumbalgia, the average pain in the leg measured 3 times a day, at predefined time points, over 4 consecutive days prior to inclusion should be more than 5 (NRS 10-point scale) 8
* Pattern of radiation suggestive for L5 or S1 pathology 49,50
* One or more positive neurological tests of nerve root tension or neurological deficit 51 ; straight leg raising test (SLRT), contralateral SLRT, motor reaction during SLRT and passive cervical flexion, motor reaction during passive cervical flexion while bending forward in standing position
* Capable of understanding the information relative to the treatment and procedure and willing to provide informed consent
* Capable of understanding and filling-out the questionnaires necessary for evaluation of the treatments
* Patients having undergone low back surgery like discectomy with or without laminectomy are allowed to participate in the study

Exclusion Criteria:

* Patients younger than 18 years
* Malignant disorder or currently under treatment for a malignant disorder
* Previous lumbar fractures
* Proven myelum lesion or abnormalities in the central neurological structures
* Systemic or connective tissue diseases
* Diabetes mellitus type I
* Multiple sclerosis
* Coagulation disorders
* Pregnancy
* Conventional medical management less then 1 month
* Pain Catastrophizing Scale > 45. When the patient has a higher score he/she will first be referred to a psychologist for consultation 52
* Leg pain due to localized hip or knee pathology
* Patients with a pacemaker or neurostimulator
* Patients previously treated with RF or PRF of the lumbar DRG

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pain reduction | 2 months

SECONDARY OUTCOMES:
Quality of life | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Maarten v Kleef, Prof. dr., Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands